CLINICAL TRIAL: NCT06204978
Title: Evaluation of Gastrointestinal Comfort Following Regular Consumption of Short-chain Fructo-oligosaccharides (10-20 g Per Day) by Children Aged 6-12 Years
Acronym: FOSTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tereos (Industry)
Collaborators: CEN Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C1712
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Gastrointestinal Tract
Keywords: ScFOS; Tolerability; Childrens
MeSH Terms: interventions — BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scFOS Dose 1 (Other): scFOS 10g
  Interventions: Dietary Supplement: short-chain fructo-oligosaccharides (dose 1); Other: Baseline
- scFOS Dose 2 (Other): scFOS 20g
  Interventions: Dietary Supplement: short-chain fructo-oligosaccharides (dose 2); Other: Baseline

INTERVENTIONS:
Dietary Supplement: short-chain fructo-oligosaccharides (dose 1) — 10 g / day at breakfast during 7 days (Day 8 - Day 14)
  Arms: scFOS Dose 1
Dietary Supplement: short-chain fructo-oligosaccharides (dose 2) — 20 g / day at breakfast during 7 days (Day 8 - Day 14)
  Arms: scFOS Dose 2
Other: Baseline — 0 g / day of short-chain fructo-oligosaccharides during 7 days (Day 1 - Day 7)

SUMMARY:
The current intake of dietary fiber by children in France and Europe is below established nutritional recommendations. Therefore, promoting fiber consumption from childhood as part of a diversified diet is crucial. For over 20 years, the food industry has been using scFOS (short-chain fructo-oligosaccharides), a fiber produced from sugar beet, as an additional source of dietary fiber. This solution can help increase daily fiber intake, meet nutritional recommendations, and provide positive health effects. Although scFOS are commonly used, there has not yet been a prospective study specifically on children aged 6 to 12 to assess gastrointestinal comfort following their regular consumption at dietary doses of 10-20 g per day.

The European Food Safety Authority (EFSA) recommends that all manufacturers document the safety of food ingredients (EFSA, 2021). This is based on Directive 2002/46/EC, which states that substances added to foods, including those intended for specific groups, must be safe and bioavailable. The study aims to assess gastrointestinal comfort and scFOS tolerance in children aged 6 to 12 and is fully compliant with Directive 2002/46/EC and EFSA recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children who were willing to participate in the study during school period;
* Have regular stool frequency: less than or equal to 3 stools per day and greater than or equal to 3 stools per week during the week prior to enrollment;
* Wanting to maintain their dietary and physical activity habits during the study;
* Agree to participate and have written informed consent from their parents or legal representatives ;
* A parent or legal representative must have a smartphone compatible with the e-PRO data collection application.

Exclusion Criteria:

* Children who had a high fiber intake, as determined by the PNNS-GS2 score during the 7 days prior to inclusion;
* Children who regularly experience gastrointestinal symptoms or have a known ongoing or chronic gastrointestinal condition;
* Children who have any known pathologies, allergies, or food intolerances;
* Children who have received antibiotic treatment in the 2 months prior to inclusion;
* Consumption of any dietary supplement or medication that affects intestinal transit or the gastrointestinal sphere (such as fiber-based supplements, prebiotics, probiotics, symbiotics, osmotic laxatives, or intestinal dressings) within the two weeks prior to inclusion;
* History of gastrointestinal tract surgery (excluding appendectomy);
* Any medical or surgical history or treatment that could potentially influence the study criteria according to the investigator;
* Children been involved in another study within the last 2 months;
* Girl who have reached menarche and experience dysmenorrhea (abdominal pain and/or changes in bowel movements);
* Parents or legal guardians who are unable to understand, speak, and read French fluently, as well as those who are likely to disregard the protocol and questionnaire completion;
* Legal representative who are unable to provide informed consent due to a court decision or any other condition that may affect their judgment;
* Not affiliated to a health insurance fund through their parents or legal representative.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal symptoms evolution | Day 1, Day 2, Day 3,…Day 14
  Daily gastrointestinal global and invidual symptom scores evaluated on 4-point Likert scales (1:none, 2:mild, 3:moderate, 4:severe) for the following symptoms: bloating, gurgling, flatulence, nausea, vomiting, abdominal pain, heartburn, acid reflux).

SECONDARY OUTCOMES:
Stool frequency evolution | Day 1, Day 2, Day 3, …Day 14
  Number of stools per day
Bristol Stool scale evolution (Stool consistency) | Day 1, Day 2, Day 3, …Day 14
  Daily score (Types 1 and 2 indicate constipation, with 3 and 4 being the ideal stools as they are easy to defecate while not containing excess liquid, 5 indicating softy stools, and 6 and 7 indicate diarrhoea)
Adverse events (except gastro-intestinal symptoms) evolution | Day 1, Day 2, Day 3, …Day 14
  Number and description of adverse event each day
Well-being evolution | Day 1, Day 2, Day 3, …Day 14
  Daily score (10-point numerical scale;from 1: "felt not at all well, in bad shape" to 10: "felt very well, in great shape");
Consumption compliance | Day 14
  Number of unused bags of product

CONTACTS AND LOCATIONS:
Locations (1):
- CEN Experimental, Dijon, Burgundy, France

IPD SHARING:
Plan to Share IPD: No